CLINICAL TRIAL: NCT04170036
Title: Do High Doses of Protein Supplements Affect Serum Lipid Profiles?
Status: Completed | Type: Observational
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Umit Yuksek, Principal Investigator, Near East University, Turkey
Other Study IDs: 2019-1-001
Record Dates: First submitted 2019-11-15; First posted 2019-11-20 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: To Study the Effects of Protein Supplements on Blood Tests
Keywords: Protein supplement; Serum creatinine; Serum sodium; Glucose metabolism; Lipid profile; C-reactive protein

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Protein supplement group: The group of subjects who use protein supplements at least for the preceding three months
  Interventions: Dietary Supplement: protein supplement
- Control group: The group of subjects who never used protein supplements

INTERVENTIONS:
Dietary Supplement: protein supplement — Protein supplement usage for at least three preceding months in varied amounts
  Groups: Protein supplement group

SUMMARY:
Protein supplements are widely used among people going to the gym. The effects of these substances on blood biochemical, hematological, inflammatuary, glucose metabolism markers and lipid profile is not well known. The previous studies on this issue give inconclusive results. So the investigators aimed to investigate this subject and compare the blood tests between subjects using and not using protein supplements.

DETAILED DESCRIPTION:
As more people are doing regular exercises, people using protein supplements are also increasing. The effects of these substances on blood lipid profiles, biochemical, hematological parameters, inflammatory and glucose metabolism markers are not well known. So the investigators of this study planned to search the effects of these substances on blood tests. Totally 69 subjects going to the gym for at least three preceding months were included to the study. They were divided into two groups: the ones using protein supplements and the ones who never used these substances. Demographic and clinical characteristics were recorded. Dietician assessed the dietary habits of the subjects. Blood was drawn for the tests mentioned above from all of the subjects. And the results were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

- Going to the gym for at least three preceding months

Exclusion Criteria:

* Any kind of acute or chronic illness
* Abnormality on electrocardiography
* Body-mass index>30 kg/m2
* Use of any kind of drugs
* Hypertension at the time of recruitment

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy population going to the gym for at least three preceding months
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Serum glucose level | 1 day
  mg/dl
Serum insulin level | 1 day
  uU/ml
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | 1 day
  No unit
Serum hemoglobine level | 1 day
  g/dl
Serum mean platelet volume | 1 day
  fL
Serum platelet level | 1 day
  x10^3/uL
Serum creatinine level | 1 day
  mg/dl
Serum urea level | 1 day
  mg/dl
Serum uric acid level | 1 day
  mg/dl
Serum aspartate aminotransferase level | 1 day
  U/L
Serum alanine aminotransferase level | 1 day
  U/L
Serum gama-glutamile transferase level | 1 day
  U/L
Serum sodium level | 1 day
  mmol/L
Serum potassium level | 1 day
  mmol/L
Serum calcium level | 1 day
  mg/dl
Serum magnesium level | 1 day
  mg/dl
Serum total cholesterol level | 1 day
  mg/dl
Serum high-density lipoprotein level | 1 day
  mg/dl
Serum low-density lipoprotein level | 1 day
  mg/dl
Serum triglyceride level | 1 day
  mg/dl
Serum C-reactive protein level | 1 day
  mg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Umit Yuksek, Dr., Principal Investigator — Near East University Cardiology Department
Locations (1):
- Near East University, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No
The subjects participated in the study do not want this.

REFERENCES:
- [Background] Salgueiro RB, Gerlinger-Romero F, Guimaraes-Ferreira L, de Castro Barbosa T, Nunes MT. Exercise training reverses the negative effects of chronic L-arginine supplementation on insulin sensitivity. Life Sci. 2017 Dec 15;191:17-23. doi: 10.1016/j.lfs.2017.10.001. Epub 2017 Oct 7. PMID 28993146